CLINICAL TRIAL: NCT02038517
Title: Insulin Secretion and Sensitivity in Subjects With Liver Cirrhosis Undergoing Orthotopic Liver Transplantation (OLT): Pre- and Post-OLT Analysis
Brief Title: Cirrhosis, Effects of TRAnsplantation and Diabetes
Acronym: CETRA
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Emanuela Orsi, MD, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Other Study IDs: EDOMP-1301
Record Dates: First submitted 2014-01-10; First posted 2014-01-16 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Liver Cirrhosis
Keywords: Insulin secretion; Insulin sensitivity; Orthotopic liver transplantation; Type 2 diabetes; Metabolic syndrome; Cardiovascular disease
MeSH Terms: conditions — Liver Cirrhosis; Insulin Resistance; Diabetes Mellitus, Type 2; Metabolic Syndrome; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Serum, plasma, urines and DNA
Oversight: Data Monitoring Committee: No

SUMMARY:
This observational study is aimed at assessing insulin secretion and sensitivity by the use of a mathematical modeling from oral glucose tolerance test in subjects with liver cirrhosis undergoing orthotopic liver transplantation (OLT), before and at various time points after OLT.

DETAILED DESCRIPTION:
Background

Diabetes is frequent in subjects with liver cirrhosis, especially in those with liver disease related to alcohol, hepatitis C, hemochromatosis and NASH, though it goes often unrecognised if screened by measuring fasting glucose. These individuals might suffer from classical type 2 diabetes, in which β-cell dysfunction plays a major role, or from hepatogenous diabetes, in which insulin resistance predominates. Orthotopic liver transplantation (OLT) improves life quality and expectancy of individuals with end-stage liver cirrhosis, thus representing the elective treatment for these patients. OLT has different effects on glucose metabolism. On the one hand, restoration of liver function reduces insulin resistance by improving hepatic insulin clearance, thus favouring regression of hepatogenous diabetes. On the other hand, OLT may worsen insulin secretion and sensitivity, due to immunosuppression and lifestyle modifications, with return to free food intake.

Aims

This observational study is aimed at assessing insulin secretion and sensitivity by the use of a mathematical modeling from oral glucose tolerance test in subjects with liver cirrhosis undergoing orthotopic liver transplantation (OLT), before and at various time points after OLT over a 10-year follow-up and to establish the relation of alterations in insulin secretion and sensitivity and their changes with transplantation with the development or persistence of abnormalities of glucose metabolism after OLT.

Secondary endpoints are to assess in these individuals:

* the relation of alterations in insulin secretion and sensitivity and their changes with transplantation with morbidity and mortality after OLT;
* the relation of alterations in insulin secretion and sensitivity and their changes with transplantation with the development or persistence of the metabolic syndrome and its components (central) obesity , dyslipidemia and hypertension;

Other pre-specified endpoints are to assess in these subjects:

* prevalence and incidence of unknown diabetes mellitus (and IFG/IGT);
* prevalence and incidence of the metabolic syndrome and its components (central) obesity , dyslipidemia and hypertension;
* morbidity and mortality from OLT-related and unrelated causes, including rejection, infection, and cardiovascular disease.

Patients Consecutive patients with normal fasting plasma glucose and HbA1c levels in waiting list for OLT will be recruited from electronic records of the diabetic clinic of the Endocrinology and Diabetes Unit, Fondazione IRCCS Cà Granda - Ospedale Maggiore Policlinico, Milan, Italy.

Measures

Routine clinical and laboratory data will be recorded at baseline and over the subsequent 10 years to obtain information about:

* cardiovascular risk factors (smoking, physical activity, family history of diabetes, dyslipidemia, hypertension and cardiovascular disease, BMI and waist circumference, total, LDL, HDL and non-HDL cholesterol, triglycerides, arterial blood pressure and HbA1c);
* cardiovascular events (myocardial infarction, stroke, lower limb ulcer/gangrene/amputation and coronary, carotid and lower limb revascularization, endovascular/surgical) and deaths.
* renal function (albumin/creatinine ratio, serum creatinine with estimation of glomerular filtration rate [eGFR]);
* current glucose-, lipid- and blood pressure-lowering and anti-platelet or anti-coagulant treatment;
* other illnesses and non-cardiovascular deaths. In addition, glucose, insulin and C-peptide levels from blood sample collected before and 15, 30, 45, 60, 90, 120', 150, and 180 min after a 75 g oral glucose tolerance test (OGTT) will be recorded. This test is routinely performed to all cirrhotic subjects before and at various time points after OLT. The response to OGTT will be evaluated by the use of a mathematical model to derive measures of insulin secretion (Proportional and Derivative Control) and sensitivity (OGIS, Oral Glucose Insulin Sensitivity).

Time schedule

This observational study was submitted for approval to the Ethics Committee of the Organization (Fondazione IRCCS Cà Granda - Ospedale Maggiore Policlinico, Milan, Italy) on October 24, 2012. The transferral of patient records (concerning the 2007-2013 visits) from the electronic database of the centre to the study database has been started on June 2013 and will terminate on September 2014.

The enrolled patients will be followed for at least 10 years with (at least) yearly visits and consultation of death records in case of drop-out for unknown reasons.

ELIGIBILITY:
Inclusion Criteria:

Subjects with end-stage liver cirrhosis in waiting list for orthotopic liver transplantation at the Fondazione IRCCS Cà Granda - Ospedale Maggiore Policlinico, Milan, Italy

Exclusion Criteria:

* Known diabetes
* Cystic fibrosis
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Secondary care outpatients clinic
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2013-06; Primary Completion 2016-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Relationship of insulin secretion and sensitivity with the development of abnormalities of glucose metabolism after OLT | 10 years
  Relation between baseline values and changes with transplantation of measures of insulin secretion and sensitivity, as derived from of the analysis of OGTT by the use of a mathematical model (i.e. proportional and derivative control for insulin secretion and oral glucose insulin sensitivity - OGIS - for insulin sensitivity ) and the development of abnormalities of glucose metabolism after OLT.

SECONDARY OUTCOMES:
Relationship of insulin secretion and sensitivity with morbidity and mortality after OLT | 10 years
  Relation between baseline values and changes with transplantation of measures of insulin secretion and sensitivity, as derived from of the analysis of OGTT by the use of a mathematical model (i.e. proportional and derivative control for insulin secretion and oral glucose insulin sensitivity - OGIS - for insulin sensitivity ) and morbidity and mortality after OLT.
Relationship of insulin secretion and sensitivity with the development of the metabolic syndrome after OLT | 10 years
  Relation between baseline values and changes with transplantation of measures of insulin secretion and sensitivity, as derived from of the analysis of OGTT by the use of a mathematical model (i.e. proportional and derivative control for insulin secretion and oral glucose insulin sensitivity - OGIS - for insulin sensitivity ) and the development of the metabolic syndrome and its components (impaired glucose metabolism, central obesity, dyslipidemia and hypertension) after OLT.

OTHER OUTCOMES:
Prevalence and incidence of impaired glucose metabolism (IFG, IGT and diabetes) | 10 years
  Prevalence of unknown diabetes mellitus or IGT (normal levels of fasting glucose and HbA1c) pre-OLT and incidence of new-onset diabetes after transplantation (NODAT) or IFG/IGT
Prevalence and incidence of the metabolic syndrome and its components (central) obesity , dyslipidemia and hypertension | 10 years
  Prevalence of the metabolic syndrome and its components (National Cholesterol Education Program - Adult Treatment Panel criteria, 2004 revision) pre-OLT and incidence of new-onset metabolic syndrome after transplantation
Morbidity and mortality after OLT | 10 years
  Morbidity and mortality from OLT-related and unrelated causes, including rejection, infection, and cardiovascular disease

CONTACTS AND LOCATIONS:
Overall Officials: Emanuela Orsi, MD, Principal Investigator — Endocrinology and Diabetes Unit, Fondazione IRCCS Cà Granda - Ospedale Maggiore Policlinico, Milan, Italy
Locations (1):
- Endocrinology and Diabetes Unit, Fondazione IRCCS Cà Granda - Ospedale Maggiore Policlinico, Milan, MI, Italy

REFERENCES:
- [Derived] Grancini V, Trombetta M, Lunati ME, Boselli ML, Gatti S, Donato MF, Palmieri E, Resi V, Pugliese G, Bonadonna RC, Orsi E. Central role of the beta-cell in driving regression of diabetes after liver transplantation in cirrhotic patients. J Hepatol. 2019 May;70(5):954-962. doi: 10.1016/j.jhep.2019.01.015. Epub 2019 Jan 21. PMID 30677460